CLINICAL TRIAL: NCT03446287
Title: Clinical Outcomes of Patients Treated With Open Surgical Repair for Complex Aortic Aneurysms
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bernardo C. Mendes, Principal Investigator, Mayo Clinic
Other Study IDs: 14-009465
Record Dates: First submitted 2018-02-21; First posted 2018-02-26 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, non-randomized, single center, data collection study of patients treated with open surgical repair (OR) for complex aortic aneurysms (CAAs).

DETAILED DESCRIPTION:
Patients in need of OR for CAAs will be placed in this prospective, non-randomized, single center, data collection study. Choice of the prosthetic graft and configuration will be based on surgeon's preference and extent of the disease. OR will be performed by vascular surgeons at Mayo Clinic, Rochester, assuming no difference in surgical techniques.

Demographics, clinical presentation, preoperative clinical and imaging assessment, intraoperative information, length of ICU stay and hospitalization, early and late mortality, major adverse events (MAEs), reintervention, rupture and QoL at different postoperative time points (4 months, 1 year, 3 years and 5 years) will be recorded according to well-designed case report forms (CRFs) and SF-36 form. Follow-up information will be obtained from office visits or mailing questionnaires (SF-36 form and CAA-specific questionnaire).

Patients will be asked to fill out the SF-36 forms preoperatively, and along with the CAA-specific questionnaire at 4 months, 1 year, 3 years and 5 years post-operatively. Physician assistants or study coordinators will interview all patients prior to treatment (during office evaluation). The follow-up assessments will be conducted by questionnaires (SF-36 and CAA-specific questionnaire) and office visits as well. If no response in 6 weeks after sending out questionnaires at each time point, telephone interview will be followed.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective, emergent or urgent OR for CAAs, including:

1. Abdominal aortic aneurysms (AAA) not eligible for endovascular aneurysm repair (EVAR), including 1) Infrarenal AAA with complex aneurysm morphology 2) Short neck infrarenal AAA 3) Juxtarenal AAA 4) Suprarenal AAA
2. Thoracoabdominal aortic aneurysms (TAAA) (Type I - IV)
3. Chronic aortic dissections

Exclusion Criteria:

1. Patients who refuse to participate the study
2. Patients age < 18 years
3. Pregnant breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open repair (OR) for complex aortic aneurysms (CAAs) at Mayo Clinic, Rochester, Minnesota will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life after open repair as measured by the Short-Form General Health Survey (SF-36) | baseline, 5 years post repair
  The SF-36 consists of 8 sub-scales which are additionally summarized into 2 summary components (physical and mental). The subscales and the summary scales both range from 0 to 100, with (0 = worst imaginable, 100 = best imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Mendes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials